CLINICAL TRIAL: NCT00703677
Title: A Pilot Trial of Lithium in Subjects With Progressive Supranuclear Palsy or Corticobasal Degeneration
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Westat (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPTUNE_PSP_CBD; HHSN265200423611C (Other Grant/Funding Number: NIH Contract)
Record Dates: First submitted 2008-06-20; First posted 2008-06-23 (Estimated); Results first posted 2010-06-11 (Estimated); Last update posted 2024-05-17 (Actual); Status verified 2024-04

CONDITIONS: Progressive Supranuclear Palsy; Corticobasal Degeneration
Keywords: progressive supranuclear palsy; corticobasal degeneration; PSP; CBD; lithium; tau
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Corticobasal Degeneration; Pick Disease of the Brain | interventions — Lithium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): All participants will receive lithium. The dosage will be titrated over a 5-week period. Participants will then be followed prospectively for 6 months. Participants will be evaluated at the screening visit, baseline visit, and weeks 2 and 5 during the titration phase. Clinic study visits will then occur on alternate months through week 28. Telephone visits will occur between clinic study visits.
  Interventions: Drug: Lithium

INTERVENTIONS:
Drug: Lithium — All participants will receive lithium. The dosage will be titrated over a 5-week period and then continued for an additional 6 months.

SUMMARY:
The goal of this trial is to evaluate the safety and tolerability of lithium in people with progressive supranuclear palsy or corticobasal degeneration.

DETAILED DESCRIPTION:
Progressive supranuclear palsy (PSP) and corticobasal degeneration (CBD) are progressive, adult-onset neurodegenerative disorders characterized by the accumulation of hyperphosphorylated tau. Symptomatic treatment is of minimal benefit to individuals with PSP or CBD, and there are no effective disease modifying agents.

Tau phosphorylation is regulated in part by the enzyme GSK-3β (glycogen synthase kinase-3 beta ). Inhibition of this enzyme may benefit individuals with PSP or CBD by decreasing the levels of phosphorylated tau. Lithium is known to inhibit GSK-3β and, thus, may be a rational therapeutic approach.

The primary objective of this study is to determine the safety and tolerability of lithium in people with PSP or CBD. Additionally, this study will evaluate potential biomarkers and clinical outcome measures as well as assess study drug compliance.

In this multicenter, open label study, 45 eligible participants with PSP or CBD will receive the study drug, lithium. The dosage of lithium will be titrated over a 5-week period, and participants will then be followed prospectively for 6 months. Participants will be evaluated at the screening visit, baseline visit, and weeks 2 and 5 during the titration phase. Clinic study visits will then occur on alternate months through week 28. Telephone visits will occur between clinic study visits.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give informed consent
2. Able to comply with the study protocol, including ability to attend follow-up study visits for the duration of the study
3. Diagnosis of PSP or CBD based on the following criteria:

   1. Probable PSP:

      * Gradually progressive akinetic disorder
      * Unequivocal and prominent slowing of vertical saccades or vertical supranuclear gaze palsy
      * Early prominent postural instability or early falls
      * Poor or absent response to levodopa
   2. Probable CBD:

      * Chronic progressive course
      * Asymmetric onset
      * Presence of higher cortical dysfunction (apraxia, apraxia of speech, non-fluent aphasia, cortical sensory loss, or alien limb)
      * Movement disorder: rigid/akinetic syndrome resistant to levodopa and either dystonic limb posturing or focal myoclonus in limb (spontaneous or stimulus sensitive)
4. If psychotropic or anti-parkinsonian medications are taken (e.g., anxiolytics, hypnotics, benzodiazepines, antidepressants, levodopa, amantadine), the dosage must be stable for 28 days prior to the screening visit and should be maintained at constant dosages throughout the study, as possible
5. If NSAIDs, ACE-Is, ARBs, thiazide diuretics, COX-2 inhibitors or theophylline are taken by the subject, the dosage must be stable for 28 days prior to the screening visit and should be maintained at constant dosages throughout the study, as possible.
6. Creatinine clearance > 50 ml/min
7. Able to take oral medication
8. Women must not be able to become pregnant (e.g., post menopausal, surgically sterile or using adequate birth control methods for the duration of the study.)
9. Able to identify a study partner

Exclusion Criteria:

1. Evidence of other diseases that could explain the clinical presentation
2. History of known sensitivity or intolerability to lithium or to other known ingredients in the study drug
3. Exposure to any investigational agent within 28 days of the screening visit
4. Clinically significant cardiac disease or EKG findings
5. Other serious illness, including psychiatric illness ("serious illness" is defined as an illness that is unstable enough that it might jeopardize the subject's ability to complete the study)
6. Moderate to severe ongoing depression
7. Family history of "PSP" or "CBS"
8. Clinically significant abnormalities on the screening visit laboratory results
9. Any AE ≥ Grade 3 as listed on the CTCAE, version 3.0
10. Women who are pregnant or breastfeeding
11. History of brain surgery
12. Use of other potential GSK-3β inhibitors (e.g., valproic acid)
13. Use of iodide salts [e.g., calcium iodide, hydrogen iodide (hydriodic acid), iodide, iodinated glycerol (Organidin), iodine, potassium iodide (SSKI), and sodium iodide]
14. Previous use of lithium
15. Use of Coenzyme Q10 at a dosage greater than 600 mg a day or NanoQuinon at a dosage greater than 150mg a day or 2.5 mg/kg a day
16. Active psoriasis

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renè Gonin, PhD, Principal Investigator — (Math. Stats.), Westat
Locations (9):
- United States (8):
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - UMDNJ Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Beth Israel Medical Center, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
- Newcastle University, Newcastle upon Tyne, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The protocol was open for recruitment between September 2008 and August 24, 2009 at neurology clinics affiliated with university hospitals.
Groups:
- Lithium Carbonate: All participants will receive lithium in this open label study (single arm). Dosages will be determined in advance to achieve serum concentrations of 0.4-0.6, 0.6-0.8, 0.8-1.0, and 1.0-1.2 mEq/L.
Period: Overall Study
Arm/Group | Lithium Carbonate
Started | 17
Completed | 14
Not Completed | 3
Not completed — Dropout-withdrawal not related to drug | 3

BASELINE CHARACTERISTICS:
Arm/Group | Lithium Carbonate
Number analyzed (Participants) | 17
Age, Customized [Number; unit: participants] — Age at enrollment
  participants
    40 - 49 years | 0
    50 - 59 years | 2
    60 - 69 years | 9
    70 - 79 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 16
  United Kingdom | 1

OUTCOME MEASURES:

1. Primary Outcome: Ability to Tolerate Lithium Carbonate
Description: The ability to complete the study period on lithium at a serum concentration of at least 0.4 mEq/L.
Time Frame: 28 weeks
Population: One subject completed the full 28 week course of study drug; 13 subjects stopped drug early due to intolerability.
Measure: Number; unit: Subject
Arm/Group | Lithium Carbonate
Number analyzed (Participants) | 14
Subject | 1

2. Secondary Outcome: Study Drug Compliance
Description: Subjects receiving 80% or more of the prescribed doses between study visits were considered compliant.
Time Frame: 28 weeks
Population: All subjects were evaluated for compliance.
Measure: Number; unit: Subjects
Arm/Group | Lithium Carbonate
Number analyzed (Participants) | 14
Subjects | 14

3. Secondary Outcome: Changes in Amount of Tau and Phosphorylated Tau in Cerebral Spinal Fluid (CSF)
Description: Progressive supranuclear palsy (PSP) and corticobasal degeneration (CBD) are characterized by hyperphosphorylation of tau. Lithium inhibits one of the kinases (GSK-3 beta) that phosphorylates tau; levels of tau phosphorylation will be measured at baseline and at Week 28.
Time Frame: 28 weeks
Population: Due to the very small number of samples collected, samples were not analyzed
Arm/Group | Lithium Carbonate
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Brain-Derived Neurotrophic Factor (BDNF) in CSF
Description: With inhibition of Glycogen Synthase Kinase (GSK)-3 beta, levels of BDNF may increase. BDNF levels will be measured at baseline and at Week 28.
Time Frame: 28 weeks
Population: Due to the very small number of samples collected, samples were not analyzed
Arm/Group | Lithium Carbonate
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in Glycogen Synthase Kinase (GSK)-3 Beta Activity
Description: Levels of beta-catenin and the ratio of phosphorylated GSK-3 beta to total GSK-3 beta will be measured at baseline and at Week 28
Time Frame: 28 weeks
Population: Due to the very small number of samples collected, samples were not analyzed.
Arm/Group | Lithium Carbonate
Number analyzed (Participants) | 0

6. Secondary Outcome: PSP Rating Scale Score: Change From Baseline
Description: The PSP Rating Scale is a 28-item scale designed to assess the disability associated with PSP. The six functional categories assessed are: daily activities, behavior, bulbar function, oculomotor function, limb motor function, and gait/midline function. Subjects will be assessed at baseline and Weeks 12, 20, and 28.
Time Frame: 28 weeks
Arm/Group | Lithium Carbonate
Number analyzed (Participants) | 0

7. Secondary Outcome: Unified Parkinson Disease Rating Scale (UPDRS) Motor Subscale Score: Change From Baseline
Description: The UPDRS is a commonly used clinical rating scale to assess motor function in patients with parkinsonism. Subjects will be assessed at baseline and Weeks 5, 12, 20, and 28.
Time Frame: 28 weeks
Arm/Group | Lithium Carbonate
Number analyzed (Participants) | 0

8. Secondary Outcome: PSP-Quality of Life Scale (QoL):Change From Baseline
Description: The PSP-QoL Scale is an instrument designed to assess mental and physical aspects of quality of life specifically in patients with PSP. Subjects will be assessed at baseline and Weeks 12, 20, and 28.
Time Frame: 28 weeks
Arm/Group | Lithium Carbonate
Number analyzed (Participants) | 0

9. Secondary Outcome: Frontal Assessment Battery (FAB): Change From Baseline
Description: The FAB is a brief, 6-item instrument designed to assess executive function. Subjects will be assessed at baseline and at Week 28.
Time Frame: 28 weeks
Arm/Group | Lithium Carbonate
Number analyzed (Participants) | 0

10. Secondary Outcome: Geriatric Depression Scale(GDS)-15:Change From Baseline
Description: The GDS-15 is a 15-item instrument used to screen for depression in the elderly. Subjects will be assessed at the Screening Visit and at Week 28.
Time Frame: 28 weeks
Arm/Group | Lithium Carbonate
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Data were collected over a 15 month period.
Description: Data were collected at scheduled clinic and telephone study visits via medical history, physical examinations, laboratory tests, EKG, and other tests as necessary. In addition, adverse events were reported to site investigators by subjects and their study partners between visits, as needed.
Arm/Group | Lithium Carbonate
Serious Adverse Events (participants affected / at risk) | 4/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithium Carbonate (N=17)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithium Carbonate (N=17)
Fatigue (General disorders) | 5 (8)
Eyelid oedema (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 4 (6)
Gait disturbance/Balance disorder (Nervous system disorders) | 9 (16)
Oedema peripheral (General disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (5)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (2)
Eye injury (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Laceration (Injury, poisoning and procedural complications) | 1 (2)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood cholesterol increased (Investigations) | 1 (1)
Blood creatine increased (Investigations) | 1 (1)
Blood glucose increased (Investigations) | 3 (3)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1)
Thyroxine increased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 3 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Posture abnormal (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Akinesia (Nervous system disorders) | 1 (1)
Aphasia (Nervous system disorders) | 1 (2)
Apraxia (Nervous system disorders) | 2 (2)
Clonus (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 3 (4)
Dysstasia (Nervous system disorders) | 2 (2)
Dystonia (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (2)
Hypokinesia (Nervous system disorders) | 4 (8)
Lethargy (Nervous system disorders) | 1 (1)
Mental impairment (Nervous system disorders) | 1 (2)
Myoclonus (Nervous system disorders) | 1 (1)
Speech disorder (Nervous system disorders) | 2 (3)
Tremor (Nervous system disorders) | 10 (13)
Cognitive deterioration (Psychiatric disorders) | 2 (2)
Confusional state (Psychiatric disorders) | 2 (2)
Depressed mood (Psychiatric disorders) | 1 (1)
Disorientation (Psychiatric disorders) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Mood altered (Psychiatric disorders) | 2 (2)
Poverty of speech (Psychiatric disorders) | 1 (1)
Social avoidant behavior (Psychiatric disorders) | 1 (1)
Staring (Psychiatric disorders) | 1 (1)
Incontinence (Renal and urinary disorders) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Activities of daily living impaired (Social circumstances) | 1 (1)
Volvulus of bowel (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The majority of subjects did not tolerate study drug, therefore, evaluations of subjects on study drug are limited in number.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Publication Policy for the National Institute of Neurological Disorders and Stroke (NINDS) Pilot Therapeutic Trials Network (NPTUNE) outlines procedures for the development and review of concept sheets, abstracts, publications, presentations. Investigators must submit an application to the NPTUNE Publications Committee for the use of data. A Writing Committee, appointed by the Publications Committee, is responsible for initiating, coordinating, and approving publications and presentations.